CLINICAL TRIAL: NCT04746573
Title: A Single Center Pilot Study to Examine the Effect of NATROX Oxygen Wound Therapy on Non-healing Wounds and the Practical Implication of Introducing a Remote Monitoring and Telehealth Solution to Manage These Complex Patients in the Home Setting.
Brief Title: Effect of Natrox Oxygen Wound Therapy on Non-healing Wounds and Implication of Remote Monitoring and Telehealth for Management in the Home.
Status: Completed | Type: Observational
Sponsor: Inotec AMD Limited (Industry)
Collaborators: Salem VA Medical Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: Inotec AMD Inc
Record Dates: First submitted 2021-01-26; First posted 2021-02-10 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Non-healing Wounds
Keywords: Diabetic foot ulcers; Venous leg ulcers; Pressure injuries; Surgical wounds
MeSH Terms: conditions — Diabetic Foot; Pressure Ulcer; Surgical Wound

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Natrox Topical Oxygen Therapy managed by telehealth: Pilot study using topical oxygen managed by telehealth in the home setting.
  Interventions: Device: Natrox Topical Oxygen Therapy

INTERVENTIONS:
Device: Natrox Topical Oxygen Therapy — Device delivering humidified oxygen directly to the wound bed

SUMMARY:
Single center pilot study examining the effect of Natrox topical oxygen therapy on chronic wounds along with the introduction of remote monitoring and telehealth for home care management.

DETAILED DESCRIPTION:
There is a wealth of evidence to support the benefits of oxygen therapy on wound healing. Oxygen is required for all major processes of wound healing and wound hypoxia is common. Skin wounds can receive oxygen from the blood stream via perfusion and from oxygen uptake through the skin. Yet, both wound perfusion and blood oxygen levels are frequently insufficient in patients with chronic wounds due to poor circulation, vascular disruption, and vasoconstriction, thereby reducing the wound's capacity to heal.

Diabetic ulcers, vascular ulcers (venous or arterial), and pressure injuries are all chronic wounds. The pathologies underlying chronic wounds can differ widely. However, common shared features include prolonged or excessive inflammation, persistent infections, and the inability to respond to reparative stimuli. Adults with vascular disease and/or diabetes are at highest risk for chronic leg and foot wounds. The ischemic (reduced tissue perfusion) and/ or hypoxic lower limb conditions which result from these conditions reduces availability of both oxygen and nutrients, making these wounds especially hard to heal. These wounds last on average 12 to 13 months, but this varies widely; many will remain open for years or never heal, and up to 30% of DFUs go onto amputation. Even when they do heal, wounds recur in 60-70% of patients, decrease quality of life, and are a significant cause of morbidity.

The need for telehealth and remote patient monitoring in the current climate is critical and reinforces the VA's strategy to protect and care for Veterans, their families, heath care providers and staff in the face of this pandemic.

The VA's tactic to shift outpatient care to a "telehealth" mode, with phone, video and/or electronic communication to meet the needs of the ambulatory patient is difficult to achieve in wound care as clinicians rely heavily on the visual appearance of the wound to direct their therapy decisions. Thus, it is imperative to validate a remote monitoring tool that offers standard telehealth care as well as accurate, consistent, and simple wound measurement and imagery. Having the ability to manage complex wounds accurately should enable quick identification of early warning signs that the wound is deteriorating thus facilitating appropriate triaging of patients that need urgent face to face medical review.

ELIGIBILITY:
Inclusion Criteria:

* Subject having non-healing wound of any etiology except for 3rd degree burns
* No visible improvement in the previous 4 weeks.
* Wound present for at least 4 weeks but less than 12 months.
* Subjects wound is not less that 1 cm sq or greater than 25 cm sq
* Subject is able and willing to participate in self care
* Subject is able and willing to follow protocol requirements
* Subject has signed informed consent

Exclusion Criteria:

* Subject has life expectancy of <1 year
* Subject is unable to manage the Natrox device.
* Subject unable or reluctant to use Iphone and imaging technology
* Subjects ulcers are 100% necrotic or if physician felt it necessary to completely cover the wound with creams or gels that would prevent the transmission of oxygen to the wound base.
* Subject has major uncontrolled medical disorder(s) such as serious cardiovascular, renal, liver or pulmonary disease, lupus, palliative care or sickle cell anemia.
* Subject is currently being treated for active malignant disease or patients with history of malignancy within the wound
* Subject has other concurrent conditions that in the opinion of the investigator may compromise subject safety
* Known contraindications to Natrox
* Known allergies to any fo the Natrox components
* Known allergies to adhesives

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with non-healing wounds of not less than 4 weeks and not greater than 12 months.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Number of participants that achieve complete wound closure. | 12 weeks
  Percentage change in ulcer size relative to baseline measurement

OTHER OUTCOMES:
Effectiveness 0f remote management and telehealth | 12 weeks
  Change in number of face to face clinic visits necessary

CONTACTS AND LOCATIONS:
Overall Officials: Dr Lee, DPM MS ABPM, Principal Investigator — US Dept of Veterans Affairs
Locations (1):
- Salem VA Healthcare, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asmis R, Qiao M, Zhao Q. Low flow oxygenation of full-excisional skin wounds on diabetic mice improves wound healing by accelerating wound closure and reepithelialization. Int Wound J. 2010 Oct;7(5):349-57. doi: 10.1111/j.1742-481X.2010.00716.x. PMID 20659184
- [Background] Babior BM. Oxygen-dependent microbial killing by phagocytes (first of two parts). N Engl J Med. 1978 Mar 23;298(12):659-68. doi: 10.1056/NEJM197803232981205. No abstract available. PMID 24176
- [Background] Knighton DR, Silver IA, Hunt TK. Regulation of wound-healing angiogenesis-effect of oxygen gradients and inspired oxygen concentration. Surgery. 1981 Aug;90(2):262-70. PMID 6166996
- [Background] 4. Lordish, H. (2000) Molecular cell biology, Freeman, New York.
- [Background] Sen CK. The general case for redox control of wound repair. Wound Repair Regen. 2003 Nov-Dec;11(6):431-8. doi: 10.1046/j.1524-475x.2003.11607.x. PMID 14617282
- [Background] Stephens FO, Hunt TK. Effect of changes in inspired oxygen and carbon dioxide tensions on wound tensile strength: an experimental study. Ann Surg. 1971 Apr;173(4):515-9. doi: 10.1097/00000658-197104000-00006. No abstract available. PMID 5573643
- [Background] Sundaresan M, Yu ZX, Ferrans VJ, Sulciner DJ, Gutkind JS, Irani K, Goldschmidt-Clermont PJ, Finkel T. Regulation of reactive-oxygen-species generation in fibroblasts by Rac1. Biochem J. 1996 Sep 1;318 ( Pt 2)(Pt 2):379-82. doi: 10.1042/bj3180379. PMID 8809022
- [Background] Frykberg RG, Banks J. Challenges in the Treatment of Chronic Wounds. Adv Wound Care (New Rochelle). 2015 Sep 1;4(9):560-582. doi: 10.1089/wound.2015.0635. PMID 26339534
- [Background] Richmond NA, Maderal AD, Vivas AC. Evidence-based management of common chronic lower extremity ulcers. Dermatol Ther. 2013 May-Jun;26(3):187-96. doi: 10.1111/dth.12051. PMID 23742279
- [Background] Stockl K, Vanderplas A, Tafesse E, Chang E. Costs of lower-extremity ulcers among patients with diabetes. Diabetes Care. 2004 Sep;27(9):2129-34. doi: 10.2337/diacare.27.9.2129. PMID 15333473

DOCUMENTS (2):
  • Study Protocol (2021-03-29): https://cdn.clinicaltrials.gov/large-docs/73/NCT04746573/Prot_001.pdf
  • Informed Consent Form (2021-04-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT04746573/ICF_002.pdf